CLINICAL TRIAL: NCT03704688
Title: A Phase 1 Trial of Trametinib and Ponatinib in Patients With KRAS Mutant Advanced Non-Small Cell Lung Cancer
Brief Title: Trial of Trametinib and Ponatinib in Patients With KRAS Mutant Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-297
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2022-02

CONDITIONS: Non Small Cell Lung Cancer; KRAS Gene Mutation
Keywords: trametinib; Ponatinib; KRAS Mutant Advanced Non-Small Cell Lung Cancer; 17-297; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trametinib; ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase I: Dose Level -3 (Experimental): Trametinib 0.5mg PO q daily Ponatinib 15mg PO q daily
  Interventions: Drug: Trametinib 0.5 mg; Drug: Ponatinib 15 MG
- Phase I: Dose Level -2 (Experimental): Trametinib 1.0 mg PO q daily Ponatinib 15mg PO q daily
  Interventions: Drug: Trametinib 1 MG; Drug: Ponatinib 15 MG
- Phase I: Dose Level -1 (Experimental): Trametinib 1.5 mg PO q daily 15mg PO q daily
  Interventions: Drug: Trametinib 1.5 MG; Drug: Ponatinib 15 MG
- Phase I: Dose Level 1 (Experimental): Trametinib 2 mg PO q daily Ponatinib 15mg PO q daily
  Interventions: Drug: Trametinib 2 mg; Drug: Ponatinib 15 MG
- Phase I: Dose Level 2 (Experimental): Trametinib 2 mg PO q daily Ponatinib 30mg PO q daily
  Interventions: Drug: Trametinib 2 mg; Drug: Ponatinib 30 MG
- Phase II (Experimental): Maximum tolerated dose as established in Phase I portion
  Interventions: Drug: Trametinib 2 mg; Drug: Ponatinib 15 MG

INTERVENTIONS:
Drug: Trametinib 0.5 mg — 0.5mg PO q daily
  Arms: Phase I: Dose Level -3
Drug: Trametinib 1 MG — 1.0 mg PO q daily
  Arms: Phase I: Dose Level -2
Drug: Trametinib 1.5 MG — 1.5mg PO q daily
  Arms: Phase I: Dose Level -1
Drug: Trametinib 2 mg — 2 mg PO q daily
  Arms: Phase I: Dose Level 1; Phase I: Dose Level 2; Phase II
Drug: Ponatinib 15 MG — 15mg PO q daily
  Arms: Phase I: Dose Level -1; Phase I: Dose Level -2; Phase I: Dose Level -3; Phase I: Dose Level 1; Phase II
Drug: Ponatinib 30 MG — 30mg PO q daily
  Arms: Phase I: Dose Level 2

SUMMARY:
The purpose of this study is to evaluate the safety of the combination of ponatinib and trametinib as well as the most appropriate dosages of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of advanced lung adenocarcinoma
* KRAS mutation
* Radiographic progression following prior treatment with platinum doublet chemotherapy and prior treatment with a PD-1/L1 inhibitor. Patients who are deemed not eligible for therapy with a PD-1/L1 inhibitor by their treating physician will also be eligible.
* Able to take oral medications
* Measurable disease as per RECIST 1.1. Previously irradiated sites of tumor may be considered measurable if there is radiographic progression at the site subsequent to the time of completing radiation.
* Karnofsky performance status (KPS) ≥ 70%
* Age >18 years old
* Adequate organ function:

  * AST, ALT ≤ 2.5 x ULN - Total bilirubin ≤ 1.5 x ULN -Albumin ≥ 2.5g/dL
  * Creatinine < 1.5 x ULN OR calculated creatinine clearance ≥ 50mL/min
  * Absolute neutrophil count (ANC) ≥ 1,200 cells/mm^3
  * Hemoglobin ≥ 9.0 g/dL
  * Platelets ≥ 100,000/mm^3
  * Amylase and lipase within normal limits (amylase ≤ 100, lipase ≤ 78)
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study drug, or
  * Agree to completely abstain from heterosexual intercourse

Exclusion Criteria:

* Patients with symptomatic brain metastasis requiring escalating doses of steroids
* Patients with grade 2 or greater diarrhea prior to study initiation despite maximal medical management
* History of acute pancreatitis within 1 year of study entry or history of chronic pancreatitis
* History of or ongoing alcohol abuse that, in the opinion of the Investigator, would compromise compliance or impart excess risks associated with study participation.
* Pregnant or lactating women
* Any type of systemic therapy (chemotherapy or experimental drugs) within 2 weeks of starting treatment on protocol
* Patients who have received prior treatment with MEK inhibitor
* A history of clinically significant interstitial lung disease or pneumonitis
* Significant uncontrolled or active cardiovascular disease, specifically including, but not restricted to: History of clinically significant (as determined by the treating physician) atrial arrhythmia; or any ventricular arrhythmia, History of congenital long QT syndrome., Abnormal QTc (≥ 450 msec in males and ≥ 470 msec in females), Ejection fraction ≤ 50% as assessed by echocardiogram.
* History of arterial thrombotic disease, specifically including, but not restricted to: Myocardial infarction or unstable angina, cerebrovascular event (CVA) or transient ischemic attack (TIA), Peripheral vascular disease or claudication.
* Uncontrolled hypertension (Diastolic blood pressure > 100 mmHg; Systolic blood pressure > 150 mmHg).
* History of venous thromboembolism (e.g. deep venous thrombosis or pulmonary embolism) within 6 months of study entry. Note: Participants enrolled after this window must be on appropriate therapeutic anticoagulation.
* History of central serous retinopathy or retinal vein occlusion
* Patients with baseline risk factors for central serous retinopathy or retinal vein occlusion such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure >21 mmHg are excluded from the trial
* History of prior malignancy within 2 years that requires treatment. Patients who are considered NED from a malignancy may be considered on a case by case basis.
* Any other condition that, in the opinion of the investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Arbour, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activity), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants were enrolled in "Phase I: Dose Level -3", "Phase I: Dose Level -2", "Phase I: Dose Level -1" and "Phase II" arms
Period: Overall Study
Arm/Group | Phase I: Dose Level -3 | Phase I: Dose Level -2 | Phase I: Dose Level -1 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Started | 0 | 0 | 0 | 7 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 7 | 5 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in "Phase I: Dose Level -3", "Phase I: Dose Level -2", "Phase I: Dose Level -1" and "Phase II" arms due to cardiovascular events observed at Dose Level 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level -3 | Phase I: Dose Level -2 | Phase I: Dose Level -1 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II | Total
Number analyzed (Participants) | 0 | 0 | 0 | 7 | 5 | 0 | 12
Age, Continuous [Median (Full Range); unit: years] |  |  |  | 58 [50 to 77] | 63 [38 to 75] |  | 61 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  | 3 | 3 |  | 6
  Male |  |  |  | 4 | 2 |  | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  |  | 0 | 1 |  | 1
  Not Hispanic or Latino |  |  |  | 7 | 4 |  | 11
  Unknown or Not Reported |  |  |  | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  | 0 | 0 |  | 0
  Asian |  |  |  | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 |  | 0
  Black or African American |  |  |  | 1 | 0 |  | 1
  White |  |  |  | 4 | 4 |  | 8
  More than one race |  |  |  | 0 | 0 |  | 0
  Unknown or Not Reported |  |  |  | 2 | 1 |  | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  |  |  | 7 | 5 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ponatinib, Phase I
Description: In the Phase I portion of the study, a standard 3+3 design will be used to find the maximum tolerated dose.
Time Frame: maximum of 18 months
Measure: Number; unit: mg of ponatinib
Groups:
- Phase I: Dose Level 1 and Dose Level 2: Dose Level 1: Trametinib 2 mg PO q daily Ponatinib 15mg PO q daily Dose Level 2: Trametinib 2mg, Ponatinib 30mg
Arm/Group | Phase I: Dose Level 1 and Dose Level 2
Number analyzed (Participants) | 12
mg of ponatinib | 30

2. Primary Outcome: Overall Response Rate
Description: In the Phase II portion of the study, RECIST criteria 1.1 will evaluate the overall response rate. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: Cardiovascular events were observed at Dose Level 2 and continued exploration of other dose levels did not proceed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level -3 | Phase I: Dose Level -2 | Phase I: Dose Level -1 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 7 | 5 | 0
Participants
  Unconfirmed Partial Response |  |  |  | 1 | 0 |
  Stable Disease |  |  |  | 4 | 2 |
  Progressive Disease |  |  |  | 0 | 1 |
  Not evaluable |  |  |  | 2 | 2 |

ADVERSE EVENTS:
Time Frame: 2 years
Description: No participants were enrolled in "Phase I: Dose Level -3", "Phase I: Dose Level -2", "Phase I: Dose Level -1" and "Phase II" arms
Arm/Group | Phase I: Dose Level -3 | Phase I: Dose Level -2 | Phase I: Dose Level -1 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 6/7 | 3/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/7 | 3/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 7/7 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level -3 (N=0) | Phase I: Dose Level -2 (N=0) | Phase I: Dose Level -1 (N=0) | Phase I: Dose Level 1 (N=7) | Phase I: Dose Level 2 (N=5) | Phase II (N=0)
Upper respiratory infection (Infections and infestations) | NA | NA | NA | NA | 2 | NA
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | NA | NA | NA | NA | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level -3 (N=0) | Phase I: Dose Level -2 (N=0) | Phase I: Dose Level -1 (N=0) | Phase I: Dose Level 1 (N=7) | Phase I: Dose Level 2 (N=5) | Phase II (N=0)
Abdominal pain (Gastrointestinal disorders) | NA | NA | NA | 2 | 0 | NA
Acute kidney injury (Renal and urinary disorders) | NA | NA | NA | 0 | 1 | NA
Alanine aminotransferase increased (Investigations) | NA | NA | NA | 0 | 1 | NA
Allergic reaction (Immune system disorders) | NA | NA | NA | 1 | 0 | NA
Alopecia (Skin and subcutaneous tissue disorders) | NA | NA | NA | 1 | 0 | NA
Anemia (Blood and lymphatic system disorders) | NA | NA | NA | 1 | 0 | NA
Anorexia (Metabolism and nutrition disorders) | NA | NA | NA | 2 | 0 | NA
Anxiety (Psychiatric disorders) | NA | NA | NA | 2 | 1 | NA
Aspartate aminotransferase increased (Investigations) | NA | NA | NA | 1 | 2 | NA
Atrial fibrillation (Cardiac disorders) | NA | NA | NA | 1 | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 1 | 1 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 1 | 0 | NA
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | NA
Chills (General disorders) | NA | NA | NA | 0 | 1 | NA
Cholesterol high (Investigations) | NA | NA | NA | 1 | 0 | NA
Constipation (Gastrointestinal disorders) | NA | NA | NA | 3 | 1 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 2 | NA
Creatinine increased (Investigations) | NA | NA | NA | 1 | 0 | NA
Delirium (Psychiatric disorders) | NA | NA | NA | 1 | 0 | NA
Diarrhea (Gastrointestinal disorders) | NA | NA | NA | 3 | 3 | NA
Dry mouth (Gastrointestinal disorders) | NA | NA | NA | 1 | 1 | NA
Dry skin (Skin and subcutaneous tissue disorders) | NA | NA | NA | 1 | 2 | NA
Dysphagia (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 4 | 3 | NA
Edema limbs (General disorders) | NA | NA | NA | 2 | 0 | NA
Ejection fraction decreased (Cardiac disorders) | NA | NA | NA | 1 | 0 | NA
Eyelid function disorder (Eye disorders) | NA | NA | NA | 1 | 0 | NA
Fatigue (General disorders) | NA | NA | NA | 2 | 0 | NA
Fever (General disorders) | NA | NA | NA | 3 | 2 | NA
Flatulence (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | NA | NA | NA | 1 | 1 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | 1 | NA
Headache (Nervous system disorders) | NA | NA | NA | 1 | 2 | NA
Heart failure (Cardiac disorders) | NA | NA | NA | 1 | 0 | NA
Hyperglycemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | NA
Hypertension (Vascular disorders) | NA | NA | NA | 3 | 1 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | NA
Hypocalcemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | NA | NA | NA | 0 | 1 | NA
Hyponatremia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | NA | NA | NA | 4 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | NA
Insomnia (Psychiatric disorders) | NA | NA | NA | 1 | 0 | NA
Lipase increased (Investigations) | NA | NA | NA | 0 | 2 | NA
Lung infection (Infections and infestations) | NA | NA | NA | 1 | 0 | NA
Lymphocyte count decreased (Investigations) | NA | NA | NA | 3 | 0 | NA
Malaise (General disorders) | NA | NA | NA | 0 | 1 | NA
Mucosal infection (Infections and infestations) | NA | NA | NA | 0 | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | 1 | NA
Myocardial infarction (Cardiac disorders) | NA | NA | NA | 0 | 1 | NA
Nausea (Gastrointestinal disorders) | NA | NA | NA | 2 | 0 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | 1 | NA
Non-cardiac chest pain (General disorders) | NA | NA | NA | 1 | 0 | NA
Oral hemorrhage (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | NA
Pain (General disorders) | NA | NA | NA | 1 | 2 | NA
Paresthesia (Nervous system disorders) | NA | NA | NA | 1 | 0 | NA
Platelet count decreased (Investigations) | NA | NA | NA | 0 | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 3 | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | NA | NA | NA | 1 | 0 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | NA | NA | NA | 5 | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | NA | NA | 4 | 1 | NA
Scalp Sensitivity (Skin and subcutaneous tissue disorders) | NA | NA | NA | 0 | 1 | NA
Serum amylase increased (Investigations) | NA | NA | NA | 0 | 1 | NA
Sinus tachycardia (Cardiac disorders) | NA | NA | NA | 1 | 0 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | NA | NA | NA | 1 | 0 | NA
Skin infection (Infections and infestations) | NA | NA | NA | 2 | 0 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 1 | NA
Supraventricular tachycardia (Cardiac disorders) | NA | NA | NA | 2 | 0 | NA
Thromboembolic event (Vascular disorders) | NA | NA | NA | 2 | 0 | NA
Upper respiratory infection (Infections and infestations) | NA | NA | NA | 0 | 1 | NA
Urinary incontinence (Renal and urinary disorders) | NA | NA | NA | 1 | 0 | NA
Urinary tract infection (Infections and infestations) | NA | NA | NA | 0 | 1 | NA
Vomiting (Gastrointestinal disorders) | NA | NA | NA | 1 | 1 | NA
Weight loss (Investigations) | NA | NA | NA | 0 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT03704688/Prot_SAP_000.pdf